CLINICAL TRIAL: NCT00164619
Title: Testing the Effectiveness of the VOICES/VOCES Intervention Package as Implemented by STD and HIV Prevention Agencies That Target Hispanics and African Americans in the U.S. and Puerto Rico
Brief Title: Testing the Effectiveness of VOICES as Implemented by STD & HIV Prevention Agencies in the US and PR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Dr. Lydia O'Donnell, Education Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4048; Contract 200-2001-00132
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Sexually Transmitted Diseases
Keywords: controlled clinical trial; behavioral intervention; prevention intervention
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Standard STD clinic services and the VOICES/VOCES intervention
  Interventions: Behavioral: VOICES/VOCES
- 2 (Active Comparator): Standard STD clinic services
  Interventions: Biological: Standard STD clinic services

INTERVENTIONS:
Behavioral: VOICES/VOCES — 45-minute intervention for small groups of African American and Hispanic heterosexual men and women. Group members are same gender and race/ethnicity. View culturally-specific condom promotion video. Facilitated group discussion to build skills in condom use and condom negotiation. Education on condom varieties to overcome participants' personal barriers to condoms use. Distribution of 3 specialty condoms of participant's choice (i.e., different sizes, textures, thicknesses, lubrication, material). [see Brief Summary above]
  Other Names: No other names
  Arms: 1
Biological: Standard STD clinic services — Individual physical exam, STD/HIV tests, treatment as indicated
  Other Names: No other names
  Arms: 2

SUMMARY:
The purpose of the project is to determine whether the VOICES/VOCES intervention, that was shown to be effective in a research study, is still effective when delivered by STD/HIV prevention agencies.

VOICES/VOCES is a brief, single-session intervention for African-American and Latino adult men and women at high risk for STD/HIV. It encourages condom use and improves condom negotiation skills. A health educator delivers the intervention to groups of 4 to 8 clinic patients in a private room. Groups are made up of people of the same sex and same race or ethnicity. Information on STD/HIV risk behaviors and condom use is delivered by culturally-specific videos, group discussion, and a poster presenting features of various condom brands. Participants role-play condom negotiation modeled in the videos. At the end of the session they are given sample condoms of their choice.

In this project, health educators from the health departments of New York City and San Juan, Puerto Rico conducted the VOICES/VOCES intervention with a sample of patients from one STD clinic in each of their cities. Researchers helped the health departments test whether the intervention is effective when local health educators deliver it.

DETAILED DESCRIPTION:
This project was an RCT with 1699 patients assigned to receive the VOICES/VOCES intervention and 1707 to receive standard of care at each of the two STD clinics (total N=3406). Participant outcomes and their measures are:

1. Change in knowledge and attitudes about condoms as determined by participant profile and survey data
2. Condom acquisition as determined by project coupon redemption data
3. STD incidence as determined by medical chart review and/or surveillance data

In addition, cost accounting data on the amounts and types of resources required to implement the intervention were used to evaluate the intervention's cost-effectiveness. Process evaluation data allow identification of factors that influenced intervention implementation and the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* STD infection at time of recruitment
* Accept treatment for STD infection at time of recruitment

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3660 (Actual)
Dates: Start 2001-07; Primary Completion 2006-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Repeat STD infection | Average of 15-months post-intervention

SECONDARY OUTCOMES:
Change in knowledge and attitudes | Immediately post-intervention
Condom coupon redemption | 3-months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lydia O'Donnell, Ed.D., Principal Investigator — Education Development Center, Inc.
Locations (2):
- Central Harlem STD Clinic, New York, New York, United States
- Centro Latino Americano de Enfermedades de Transmission Sexual, San Juan, Puerto Rico

REFERENCES:
- [Background] O'Donnell CR, O'Donnell L, San Doval A, Duran R, Labes K. Reductions in STD infections subsequent to an STD clinic visit. Using video-based patient education to supplement provider interactions. Sex Transm Dis. 1998 Mar;25(3):161-8. doi: 10.1097/00007435-199803000-00010. PMID 9524995